CLINICAL TRIAL: NCT01608828
Title: Assessing the Functional and Psychosocial Impact of Strabismus in Asian Children Using the AS-20 and IXTQ Questionnaires
Status: Completed | Type: Observational
Sponsor: Singapore National Eye Centre (Other Government)
Responsible Party: Principal Investigator, Audrey Wei-Lin Chia, Senior Consultant, Singapore National Eye Centre
Other Study IDs: 2012/350/A
Record Dates: First submitted 2012-05-28; First posted 2012-05-31 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Strabismus
MeSH Terms: conditions — Strabismus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Studies suggest that strabismus has a negative impact on a person's self-image, interpersonal relationships, emotional and psychosocial state (4-15). There are, however, few such studies based in Asia, and the functional and psycho-social impact of disease is often neglected in our management of strabismus in Singapore. The aim of this pilot study is to measure quality-of-life (QOL) among strabismic children in Singapore so as to better understand the functional and psychosocial issues faced by these children in their daily living. The investigators also hope to evaluate the performance of the Intermittent Exotropia Questionnaire (IXTQ) (2) and Adult Strabismus Quality of Life Questionnaire (AS-20) (1) and to determine if differences between child and parental perceptions exist.

60 children with strabismus presenting to the KKWCH Eye Centre and their parents will be invited to participate in the study and answer questions in 2 Pediatric Eye Disease Investigator Group (PEDIG)-validated questionnaires (i.e. the IXTQ and AS-20). 30 children aged 5-7 years will answer the 12-question IXTQ (5-7 years), while 30 children aged 8-16 years will answer the 12-question IXTQ (8-16 years) and the 20-question AS-20 questionnaires. Their parents will answer the self-administered IXTQ child-proxy (12 questions), IXTQ parental (17 questions) and modified AS20 child-proxy questionnaires (20 questions). For comparison, 60 aged-matched children without strabismus or amblyopia (30 aged 5-7 years, and 30 aged 8-16) and their parents will also be invited to answer similar questionnaires (controls).

Results will be analysed question-by-question and then by composite score, and comparison will be made between child and parental-proxy measures, as well as with scores obtained from myopic children. It is hoped, that from this study, we will be able to assess the usefulness of the IXTQ and AS-20 instruments as measures of QOL in strabismic children, and to assess the feasibility of its use in a larger study looking at the impact of strabismus and its treatment in Singaporean children.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 5 to 16 years (inclusive) with strabismus or age-matched controls without strabismus/amblyopia
2. Any tropia
3. Willingness of children or parents willing to complete questionnaires
4. Parents with sufficient reading skills to complete the English written IXTQ and AS20
5. Parent/guardian able to provide informed consent

Exclusion Criteria:

1. Children with poor vision (VA worse than 6/7.5) in either eye
2. Children with any ocular, neurological or syndromic problems
3. Children with developmental delay or mental impairment
4. Children from overseas (not residing in Singapore)

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with strabismus
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Quality of life in Asian children with strabismus | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- KK Women and Children Hospital, Singapore, Singapore